CLINICAL TRIAL: NCT02435550
Title: iCare for Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Halted due to funding issues.
Sponsor: University of Florida (Other)
Collaborators: Cellworks Group Inc. (Industry); Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB201500073; OCR14209 (Other: OnCore)
Record Dates: First submitted 2015-04-20; First posted 2015-05-06 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia; Acute Myelogenous Leukemia; Acute Lymphoid Leukemia; Leukemia, Acute Lymphoblastic; Multiple Myeloma; Myelofibrosis
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Multiple Myeloma; Primary Myelofibrosis | interventions — Molecular Diagnostic Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Acute Myeloid Leukemia (Experimental): Patients with acute myeloid leukemia will have blood, bone marrow aspirate, and saliva collected from them as part of routine care.
  Interventions: Genetic: Molecular diagnostic testing
- Acute Lymphoblastic Leukemia (Experimental): Patients with acute lymphoblastic leukemia will have blood, bone marrow aspirate , and saliva collected from them as part of routine care.
  Interventions: Genetic: Molecular diagnostic testing
- Myelodysplastic Syndrome (Experimental): Patients with myeloplastic syndrome will have blood, bone marrow aspirate, and saliva collected from them as part of routine care.
  Interventions: Genetic: Molecular diagnostic testing
- Myelofibrosis (Experimental): Patients with myelofibrosis will have blood, bone marrow aspirate, and saliva collected from them as part of routine care.
  Interventions: Genetic: Molecular diagnostic testing
- Multiple Myeloma (Experimental): Patients with multiple myeloma will have blood, bone marrow aspirate, and saliva collected from them as part of routine care.
  Interventions: Genetic: Molecular diagnostic testing

INTERVENTIONS:
Genetic: Molecular diagnostic testing — Molecular diagnostic testing will be performed on peripheral blood, bone marrow aspirate and saliva samples that will be collected from each patient as part of routine care. Tests performed may include: cytogenetics, FISH, chromosome copy number variation, next generation DNA sequencing, methylation, and metabolomics.

SUMMARY:
The purpose of this study is to use genomic information from individual patients to create simulation avatars that will be used to predict novel drug combinations with therapeutic potential.

DETAILED DESCRIPTION:
As part of normal clinical care, subjects will undergo peripheral blood draws and biopsies for disease assessment of their cancer. In cases of hematological malignancies, bone marrow aspiration & biopsy are routinely performed.

As part of this project, the following will be done to the samples collected and with clinical outcomes data:

* donate peripheral blood specimens whenever blood is already being drawn for clinical purposes.
* donate bone marrow aspiration samples whenever a bone marrow aspiration procedure is already being done for clinical purposes.
* donate saliva whenever blood draw is already being done for clinical purposes.
* allow the investigators to perform gene mutation profiling.
* allow the investigators to study gene mutation results.
* allow the investigators to perform pharmacogenetic profiling.
* allow the investigators to study pharmacogenetic profiles.
* allow the investigators to examine chromosome copy number variations.
* allow the investigators to examine genomic methylation.
* allow the investigators to quantify metabolomics/cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Individuals known or suspected of having a blood cancer or hematologic disorder
* Individuals with presence of extramedullary disease
* Capable of providing informed consent.

Exclusion Criteria:

* Does not have a blood cancer or a hematologic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Overall Response | Up to 5 years
  The overall response rate (ORR) is defined as achieving a complete remission (CR), partial remission (PR), and/or hematological improvement based on 2006 International Working Group (IWG) criteria (Cheson, et al. Blood 2006).

SECONDARY OUTCOMES:
Number of patients with drug-related Grade 3 and Grade 4 adverse events | Up to 5 years
  Toxicity will be assessed by the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) v 4. Adverse event incidences will be compared to individual pharmacogenetic gene variants.
Progression-free survival after treatment | Up to five years
  The disease free survival will be analyzed using Kaplan-Meier method and comparisons made to computer predicted response.
Overall survival after treatment | Up to 5 years
  The overall survival will be analyzed using Kaplan-Meier method and comparisons made to computer predicted response.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R. Cogle, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Shands Cancer Hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No